CLINICAL TRIAL: NCT06737185
Title: Comparison of Speech Understanding Between Tonotopy-based Fitting and Evolutionary Algorithm-based Setting: a Prospective Cross-sectional Study
Brief Title: Comparison of Speech Understanding Between Tonotopy-based Fitting and Setting Based on Evolutionary Algorithms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MEDEL_algoevIC_Dijon_study
Record Dates: First submitted 2024-12-05; First posted 2024-12-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant; evolutionary algorithms; tonotopy-based fitting
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EA arm (Other): at 6 month post-activation: evolutionary algorithms to modify the tonotopy-based fitting FS4T to give EAFS4T fitting.
  Participant wears EAFS4T during 6 weeks.
  Interventions: Other: EAFS4T: modification with evolutionary algorithm of tonotopic-based fitting

INTERVENTIONS:
Other: EAFS4T: modification with evolutionary algorithm of tonotopic-based fitting — Comparison of FS4T and EAFS4T
  Other Names: FS4T: tonotopic-based fitting

SUMMARY:
Main objective:

Compare speech recognition in noise with tonotopic setting (FS4T) and with tonotopic fitting modified by evolutionary algorithm (EAFS4T) in adult patients implanted for 6 months or more with a MED-EL cochlear implant with FS4T.

Secondary objectives:

Comparison of FS4T and EAFS4T settings

* for speech recognition in quiet
* for subjective auditory spatial perception
* for subjective auditory and musical perception

DETAILED DESCRIPTION:
Introduction: Cochlear implantation allows the rehabilitation of profound bilateral deafness, restoring speech perception and verbal communication when the traditional hearing aid no longer provides satisfactory hearing gain. A cochlear implant includes an electrode array and its functioning is based on the principle of cochlear tonotopy: each electrode encodes a frequency spectrum according to its position in the cochlea (high frequencies are assigned to the basal electrodes and low frequencies to the apical electrodes). The cochlear implant thus breaks down the frequency spectrum into a number of frequency bands via bandpass filters corresponding to the number of electrodes in the implant. During the fitting these bands can be modified by the audiologist. The fitting software developed by the manufacturers proposed a default fitting with a lower limit between 100 and 250 Hz according to the brands and an upper limit of about 8500 Hz. The frequency bands assigned to each electrode follow a logarithmic scale with the high frequencies for the basal electrodes and the low frequencies for the apical electrodes. This distribution takes into account the number of active electrodes but does not take into account the anatomy and the natural cochlear tonotopy specific to each patient. Several studies have analyzed the anatomical variations of the cochlear dimensions: size of the cochlea and the ratio between the contact surfaces of the electrodes with the cochlea are variable from one patient to another. The insertion depth during surgery is also variable due to parameters related to the patients as well as to the operator, which seems to impact the understanding of speech in noise. Mathematical algorithms have recently been developed to estimate the cochlear tonotopy of each patient from a CT scan assessment. CT imaging of the implanted ear combined with 3D reconstruction software, provides cochlear length measurements Using this approach it is possible to measure the position of each electrode relative to the cochlear apex. Recently, MED-EL (Austria) has developed a new approach based on CT-scan and tuning of the frequencies associated with each electrode using anatomical information of position of the electrodes in the cochlea: this fitting is called anatomy-based fitting.

A tonotopy-based fitting allows for better results in pitch perception or speech perception in noise or musical perception. However, there is a large variability in the results observed between patients. This variability could be due to the individual characteristics of the listeners (neuronal survival, current propagation and spread, duration of deafness, lack of cortical plasticity).

A modification of frequency allocations in the setting could take into account this individual variability and improve speech discrimination and music perception. Saadoun et al. (2022) studied on 27 subjects the effect of an adjustment of frequency allocation by an evolutionary algorithm (EA) approach and showed an improvement in speech perception in noise compared to a default setting (not based on tonotopy) for patients implanted for more than 6 months in a bimodal situation (with a contralateral prosthesis). We therefore propose to use evolutionary algorithms to modify the tonotopy-based fitting and improve the perception in noise of implanted patients.

Main objective:

Compare speech recognition in noise with tonotopic setting (FS4T) and tonotopic fitting modified by evolutionary algorithm (EAFS4T) in adult patients implanted for 6 months or more with a MED-EL cochlear implant with FS4T.

Secondary objectives:

Comparison of FS4T and EAFS4T settings

* for speech recognition in quiet
* for subjective auditory spatial perception
* for subjective auditory and musical perception

Plan of the study: It is a prospective open monocentric transversal study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>= 18 years old) speaking French
* Patient who fulfils the criteria for cochlear implantation

Exclusion Criteria:

* retro-cochlear pathology: auditory neuropathy, vestibular schwannoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Speech recognition in noise | 6 weeks after EAFS4T fitting
  HINT-5 min test. Noise level: 60 dB SPL. Speech level: adaptive with the answers of the participant. Result: speech-to-noise ratio (speech reception threshold, SRT50) for 50% of intelligibility in noise.
  Test with EAFS4T and with FS4T.

SECONDARY OUTCOMES:
Speech recognition in quiet | 6 weeks after EAFS4T fitting
  One list of 10 disyllabic words (Fournier lists) at 65 dB SPL. The participant has to repeat the word emitted.
  Result: score on 10. Test with EAFS4T and with FS4T
Subjective auditory spatial perception | at EAFS4T fitting (6 months after cochlear implant activation) and 6 weeks after EAFS4T fitting
  SSQi15 questionnaire (" Speech, Spatial, and Qualities of hearing scale ", SSQ). The questionnaire consists of 15 questions describing various real-world hearing situations.
  The subject answers each question with a score on a visual analogue scale graduated from 0 to 10 ranging from "not at all" to "yes perfectly".
  The result obtained is composed of
  * a total average score equal to the sum of the scores of all the questions divided by the total number of questions.
  * 3 average sub-scores describing 3 subscales: Speech hearing with 5 questions, Spatial hearing with 5 questions, Quality of hearing with 5 questions.
  Questionnaire with FS4T (at EAFS4T fitting) and with EAFS4T (6 weeks after EAFS4T fitting)
Subjective assessment of auditory perception | at EAFS4T fitting (6 months after cochlear implant activation) and 6 weeks after EAFS4T fitting
  Assessment of sound quality in silence and in noise with 4 statements. Likert scale from 1 to 5. Score on 20.
  Likert scale with FS4T (at EAFS4T fitting) and with EAFS4T (6 weeks after EAFS4T fitting)
Subjective assessment of musical perception | at EAFS4T fitting (6 months after cochlear implant activation) and 6 weeks after EAFS4T fitting
  Six questions from the Munich Music Self-Questionnaire [Stark et al. 2003]. Questionnaire with FS4T (at EAFS4T fitting) and with EAFS4T (6 weeks after EAFS4T fitting)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis BOZORG GRAYELI, Pr, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (1):
- CHU, Dijon, France

IPD SHARING:
Plan to Share IPD: No